CLINICAL TRIAL: NCT06668831
Title: Fibroblast Growth Factor 23 and Risk of Cardiac Arrhythmias in Hemodialysis Patients: a Proof-of-concept Study (FibCa-HD)
Brief Title: Fibroblast Growth Factor 23 and Risk of Cardiac Arrhythmias in Hemodialysis Patients
Acronym: FibCA-HD
Status: Recruiting | Type: Observational
Sponsor: Antonio Bellasi (Other)
Responsible Party: Sponsor-Investigator, Antonio Bellasi, Nephrology Consultant and Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: FibCA-HD
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis
Keywords: fgf23; cardiac arrhythmia; QTc; cardiovascular risk
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All study biological materials (serum sample) will be stored in the EOC biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects on maintenance hemodialysis: The study envisages the enrolment of:
  * adult subjects (>18 years of age) who are able to sign an informed consent.
  * on maintenance HD (for at least 3 months)
  * without history of cardiac arrhythmias at study recruitment define as atrial fibrillation or pace-maker assisted cardiac rhythm

SUMMARY:
Despite recent progress in the field of hemodialysis (HD), mortality remains unacceptably high, particularly due to cardiac arrhythmias. Recent evidence suggests that fibroblast growth factor 23 (FGF23) is implicated in the pathogenesis of cardiac arrhythmias and sudden death. However, several aspects of both the pathogenetic mechanism(s) as well as the actual association in individuals with Chronic Kidney Disease (CKD) and the effect of dialysis clearance of FGF23 need to be elucidated.

The investigators aim at testing the independent association of FGF23 changes due to dialysis removal and electrocardiographic (ECG) abnormalities (namely QTc prolongation) in a well characterized sample of patients undergoing maintenance HD. The study will be developed in the Division of Nephrology, Ente Ospedaliero Cantonale.

DETAILED DESCRIPTION:
This is an exploratory, observational, prospective, mono-center study that aims to elucidate the pathogenesis of cardiac repolarization and arrhythmias in subjects with CKD receiving maintenance dialysis.

This exploratory research project aims to confirm the link between FGF23 and ECG abnormalities (QTc as a proxy for cardiac arrhythmias) in a well-characterized sample of HD patients and expand our understanding of the molecular mechanisms by which FGF23 may trigger arrhythmias.

Previous works suggest that FGF23 cardiac toxicity may be mediated by the activation of FGFR4 and that modulation of FGF23-FGFR4 signaling through monoclonal antibodies can attenuate the toxic effects of FGF23 on the CM. Although these preliminary data warrant clinical and molecular confirmation, they also suggest FGF23-FGFR4 modulation as a novel potential therapeutic target in CKD to improve morbidity and mortality.

During a standard dialysis session, FGF23 is acutely removed while Ca2+ is provided to the patients. However, shortly after the HD session completion, it was documented that FGF23 serum levels rebound. The investigators hypothesize that acute reduction and subsequent rebound of circulatory levels of FGF23 coupled with calcium loading induced by HD may favour a Ca 2+ influx in the CM and trigger cardiac arrhythmias.

This exploratory study aims to determine the independent association between variations in serum levels of FGF23 and QTc (msec) during and after dialysis. In particular, the primary endpoint of the study is defined as the association between QTc variations (msec) defined as the difference between QTc pre-dialysis and QTc 1 hour after dialysis session completion and variations of serum levels of FGF23 defined as the difference between serum levels of FGF23 at dialysis session completion and after 1-hour form dialysis session completion. The investigators hypothesize that these time points should maximize the chance of detecting a significant association between the exposure variable (FGF23) and the outcome of interest (QTc).

All study procedures are non-invasive, and they will be carried out between the beginning of the last HD of the week and the beginning of the first HD of the following week (long interdialytic interval) to allow for the maximum variation of serum levels of FGF23 between dialysis sessions.

All study-related procedures are performed on top of standard clinical practice, and guidelines are performed non-invasively. Study participants will undergo the following procedures:

* ECG: A standard 12-leads ECG will be recorded at the beginning, at the end as well as 60 minutes after the end of the last HD session of the week and at the beginning of the first HD session of the following week. All readings will be performed will be centralized and read by a single investigator blinded to clinical information at EOC.
* Laboratory assessment: a blood sample will be taken at the beginning, at the end, and 60 minutes after the end of the last HD session of the week and at the beginning of the first HD session of the following week. Laboratory investigations will check the serum values of cardiovascular biomarkers (including FGF23) associated with QTc and volume expansion (OH: overhydration). Venous blood samples for measurement of cardiovascular biomarkers will be drawn at each time point and stored in the biobank at Ente Ospedaliero Cantonale (EOC) according to the standard procedures. These aliquotes will be used to assess FGF23 and for subsequent in-vitro evaluation of the cardiac arrhythmogenicity of patients' sera in relation to the homeostasis variation induced by HD.
* Volume assessment: total body weight will be measured at dialysis session, to calculate the net body weight increase during the long interval. Overhydration (OH) will be quantitatively assessed with a portable whole-body bioimpedance spectroscopy device (Fresenius Medical Care GmbH, Bad Homburg, Germany). The total body water (TBW), the extracellular water (ECW), the intracellular water (ICW), and the OH are calculated as previously defined
* Applanation tonometry: Central blood pressure (BP) values and aortic pressure waveforms will be obtained non-invasively directly from the common carotid artery using a validated high fidelity PulsePen tonometer (DiaTecne, San Donato Milanese, Italy). In particular, the subendocardial viability ratio (SEVR) will be calculated during the first HD session of the week according to the central BP wave form as previously reported
* Echocardiogram: If no echocardiogram exam within 12 months from study inception is available in the patient's chart, a two-dimensional echocardiographic study will be performed before the first HD session of the week utilizing a standard equipment as per standard clinical practice. Digital images will be acquired in the long axis and short axis parasternal views and the apical four and two chamber views and three-cycle clips will be stored on magnetic optical disks for future review. The presence of valvular calcification (aortic and mitral valve) as well as systolic and diastolic function assessment will be performed.

Adverse event: The occurrence of any adverse events (AE) will be recorded for the occurrence of any event from study inception until the end of the following week This exploratory study will be carried out at the Division of Nephrology, Ente Ospedaliero Cantonale (EOC), Ticino, Switzerland.

ELIGIBILITY:
The study envisages the enrolment of:

* Adult subjects (>18 years of age) who can sign an informed consent.
* on maintenance HD (for at least 3 months)

Exclusion Criteria:

* history of cardiac arrhythmias at study recruitment define as atrial fibrillation or pace-maker assisted cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects on maintenance hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Associations of QTc and FGF23 changes | the primary endpoint will be assessed one hour after dialysis cessation
  The primary endpoint of the study is defined as the association between QTc variations (msec) defined as a continuous variable as the difference between QTc pre-dialysis and QTc 1 hour after dialysis session completion and variations of serum levels of FGF23 defined as a continuous variable as the difference between serum levels of FGF23 at dialysis session completion and after 1-hour form dialysis session completion. We hypothesize that these time points should maximize the chance of detecting a significant association between the exposure variable (FGF23) and the outcome of interest (QTc).

SECONDARY OUTCOMES:
To gauge the dynamic association between FGF23 and QTc we will also explore | these endpoints will be assessed between dialysis session initiation and 1 hour after dialysis session cessation
  A. Association of serum levels of FGF23 and QTc (msec) at dialysis session initiation (both utilized as continuous variables) B. Association of serum levels of FGF23 and QTc (msec) at dialysis session completion C. Association of serum levels of FGF23 and QTc (msec) 1 hour after dialysis session completion D. Association of QTc variations (msec - defined as the difference between QTc pre-dialysis and QTc after dialysis session completion) and serum levels of FGF23 variations before and after dialysis session completion (defined as the difference between serum levels of FGF23 at dialysis session initiation and dialysis session completion) E. Association of QTc variations (msec - defined as the difference between QTc at dialysis session completion and QTc 1 hour after dialysis session completion) and serum levels of FGF23 variations before and 1 hour after dialysis session completion (defined as variable as the difference between serum levels of FGF23 at dialysis session completion)
To gauge the dynamic association between FGF23 and QTc we will also explore | These endpoints will be assessed bewteen the beginning of the last dialysis of the week and the beginning of the first dialysis of the following week (72 hours)
  A. Association of QTc variations (msec - defined as the difference between QTc at dialysis session completion and QTc 72 hours after dialysis session completion) and serum levels of FGF23 variations before and after 72 hours from dialysis session completion (defined as the difference between serum levels of FGF23 at dialysis session completion and 72 hours after dialysis session completion).
  B. Association of serum levels of FGF23 and QTc (msec) at the beginning of the first dialysis of the week, after the long interdialytic interval.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Bellasi, MD, PhD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Servizio di Nefrologia, Ospedale Regionale di Lugano, Civico, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
IPD maybe shared upon request and in respect with the regulation on data protection

REFERENCES:
- [Background] Arrigo M, Von Moos S, Gerritsen K, Sadoune M, Tangvoraphonkchai K, Davenport A, Mebazaa A, Segerer S, Cippa PE. Soluble CD146 and B-type natriuretic peptide dissect overhydration into functional components of prognostic relevance in haemodialysis patients. Nephrol Dial Transplant. 2018 Nov 1;33(11):2035-2042. doi: 10.1093/ndt/gfy113. PMID 29733422
- [Background] Tiong MK, Krishnasamy R, Smith ER, Hutchison CA, Ryan EG, Pascoe EM, Hawley CM, Hewitson TD, Jardine MJ, Roberts MA, Cho Y, Wong MG, Heath A, Nelson CL, Sen S, Mount PF, Vergara LA, Paul-Brent PA, Johnson DW, Toussaint ND. Effect of a medium cut-off dialyzer on protein-bound uremic toxins and mineral metabolism markers in patients on hemodialysis. Hemodial Int. 2021 Jul;25(3):322-332. doi: 10.1111/hdi.12924. Epub 2021 Mar 28. PMID 33779046
- [Background] Fu X, Cui QQ, Ning JP, Fu SS, Liao XH. High-Flux Hemodialysis Benefits Hemodialysis Patients by Reducing Serum FGF-23 Levels and Reducing Vascular Calcification. Med Sci Monit. 2015 Nov 11;21:3467-73. doi: 10.12659/msm.894894. PMID 26558428
- [Background] Sikaneta T, Ho N, Bellasi A, Mahdavi S, Taskapan H, Svendrovski A, Makanjee B, Roberts J, Wu G, Nathoo B, Tam P. QTc Interval Prolongation Is Independently Associated with FGF23 and Predicts Mortality in Predialysis Chronic Kidney Disease. Cardiorenal Med. 2024;14(1):45-57. doi: 10.1159/000535133. Epub 2024 Jan 8. PMID 37963445
- [Background] Graves JM, Vallejo JA, Hamill CS, Wang D, Ahuja R, Patel S, Faul C, Wacker MJ. Fibroblast growth factor 23 (FGF23) induces ventricular arrhythmias and prolongs QTc interval in mice in an FGF receptor 4-dependent manner. Am J Physiol Heart Circ Physiol. 2021 Jun 1;320(6):H2283-H2294. doi: 10.1152/ajpheart.00798.2020. Epub 2021 Apr 30. PMID 33929896
- [Background] Di Iorio B, Bellasi A. QT interval in CKD and haemodialysis patients. Clin Kidney J. 2013 Apr;6(2):137-43. doi: 10.1093/ckj/sfs183. Epub 2013 Jan 17. PMID 26019841
- [Background] Vazquez-Sanchez S, Poveda J, Navarro-Garcia JA, Gonzalez-Lafuente L, Rodriguez-Sanchez E, Ruilope LM, Ruiz-Hurtado G. An Overview of FGF-23 as a Novel Candidate Biomarker of Cardiovascular Risk. Front Physiol. 2021 Mar 9;12:632260. doi: 10.3389/fphys.2021.632260. eCollection 2021. PMID 33767635
- [Background] Niu J, Shah MK, Perez JJ, Airy M, Navaneethan SD, Turakhia MP, Chang TI, Winkelmayer WC. Dialysis Modality and Incident Atrial Fibrillation in Older Patients With ESRD. Am J Kidney Dis. 2019 Mar;73(3):324-331. doi: 10.1053/j.ajkd.2018.09.011. Epub 2018 Nov 16. PMID 30449517
- [Background] Rantanen JM, Riahi S, Schmidt EB, Johansen MB, Sogaard P, Christensen JH. Arrhythmias in Patients on Maintenance Dialysis: A Cross-sectional Study. Am J Kidney Dis. 2020 Feb;75(2):214-224. doi: 10.1053/j.ajkd.2019.06.012. Epub 2019 Sep 18. PMID 31542235
- [Background] Di Lullo L, Rivera R, Barbera V, Bellasi A, Cozzolino M, Russo D, De Pascalis A, Banerjee D, Floccari F, Ronco C. Sudden cardiac death and chronic kidney disease: From pathophysiology to treatment strategies. Int J Cardiol. 2016 Aug 15;217:16-27. doi: 10.1016/j.ijcard.2016.04.170. Epub 2016 May 3. PMID 27174593
- See also: STROBE statement — http://www.jclinepi.com/article/S0895-4356(07)00436-2/pdf
- See also: Declaration of Helsinki — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects
- See also: Ordinance on Human Research with the Exception of Clinical trials (HRO) — https://www.admin.ch/opc/en/classified-compilation/20121177/index.html
- See also: Human Research Act (HRA) — http://www.admin.ch/opc/en/classified-compilation/20121176/201401010000/810.305.pdf